CLINICAL TRIAL: NCT03779984
Title: Use of a Red-Rubber Catheter to Facilitate Nasotracheal Intubation in Adult Patients: A Prospective Randomized Controlled Trial
Brief Title: Red-Rubber Catheter to Facilitate Nasotracheal Intubation in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, David W Mercier, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: STU-2018-0190
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome accessor and participants are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Red Rubber Catheter Group (Experimental): Red Rubber Catheter (RRC) guided nasal tracheal intubation; a RRC securely attached to nasal tracheal tube and the rounded end of the catheter introduced into a naris.
  Interventions: Device: Red Rubber Catheter
- Standard nasal tracheal intubation (Sham Comparator): The nasotracheal tube will be inserted into the nasal passage.
  Interventions: Device: Standard nasal tracheal Intubation

INTERVENTIONS:
Device: Red Rubber Catheter — Experimental group will be intubated with red rubber catheter guidance
  Arms: Red Rubber Catheter Group
Device: Standard nasal tracheal Intubation — Control group will be intubated with standard nasal tracheal tube without guidance
  Other Names: Nasal tracheal intubation without guidance
  Arms: Standard nasal tracheal intubation

SUMMARY:
This study was designed to compare the effectiveness of using a red-rubber catheter versus standard, direct insertion of a thermosoftened, lubricated nasal endotracheal tube into the naris to facilitate nasotracheal intubation in adults. This study will assess if the red-rubber catheter method leads to lower incidence and severity of epistaxis, faster time to intubation, and higher patient satisfaction compared to the current standard of care.

DETAILED DESCRIPTION:
The study population for this prospective randomized controlled trial will consist of male and female adult subjects over the age of 18 having surgery requiring nasal tracheal intubation (NTI). Subjects will be randomized to either the Red Rubber Catheter (RRC) group or control group.

Oxymetazoline nasal spray will be administered with 1 spray per nostril preoperatively. Premedication with glycopyrrolate 0.2 mg and benzodiazepine at discretion of provider will be given preoperatively. Subjects will then be brought into the operating room and placed on all standard ASA monitors (BP cuff, EKG, pulse oximetry). One spray of oxymetazoline per nostril will again be administered. Standard preoxygenation will be used with a face mask and 100% O2. After induction of anesthesia, provider will confirm mask ventilation and 1 more spray of oxymetazoline will be administered per nostril. Intubation will first be attempted via a naris. Size 6.5 nasotracheal RAE tubes (Shiley Nasal RAE Tracheal Tube with TaperGuard Cuff, manufactured by Coviden llc, Mansfield, MA 02048) will be used in female patients and size 7.5 in males. The tubes will be thermosoftened by allowing them to sit in warm saline prior to use. Water-based lubrication will be used for dilation and intubation. Time from insertion of RRC or NETT into nasal passage to first recording of end-tidal CO2 will be recorded. Direct video laryngoscopy will be used to facilitate placement of the nasotracheal RAE tube.

Five minutes after intubation, a non-collaborating anesthesia provider blinded to the method of intubation will grade the severity of bleeding by performing direct video laryngoscopy, inspecting the posterior pharynx and using a scale -

1. No epistaxis (no blood observed on either the surface of the tube or the posterior pharyngeal wall);
2. Mild epistaxis (blood apparent on the surface of the tube or posterior pharyngeal wall);
3. Moderate epistaxis (pooling of blood on the posterior pharyngeal wall);
4. Severe epistaxis (a large amount of blood in the pharynx impeding nasotracheal intubation-before the epistaxis assessor enters the operating room, requiring suction for intubation or necessitating urgent orotracheal intubation.)

Degree of patient satisfaction and nasal pain on the side of intubation will be rated on a numerical rating scale at 30 and 60 minutes in the post-anesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, male and female
* Subjects undergoing surgery requiring NTI
* ASA 1-3

Exclusion Criteria:

* History of anticoagulant use or coagulopathy
* History of latex allergy
* History of difficult airway
* Anticipated difficult airway requiring awake intubation
* Abnormal anatomy of the nasal passage (due to prior trauma, surgery, congenital defects, etc.) or basilar skull fracture
* Patients unable to be placed in the sniffing position
* Morbid obesity with BMI > 40
* Pregnancy
* ASA 4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Riccio, MD, Study Director — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Heath Hospital System, Dallas, Texas
  - MD Anderson Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Red Rubber Catheter Group | Standard Nasal Tracheal Intubation
Started | 56 | 56
Completed | 56 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 112 participants enrolled to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Red Rubber Catheter Group | Standard Nasal Tracheal Intubation | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.37 (16.50) | 56.75 (16.26) | 57.06 (16.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 35 | 34 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 56 | 56 | 112
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 27.28 (5.01) | 26.33 (4.90) | 26.81 (4.95)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Nasal Bleeding
Description: The number of participants with nasal bleeding within 5 minutes following nasal tube placement.
Time Frame: Within 5 minutes following the nasal tracheal intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Red Rubber Catheter Group | Standard Nasal Tracheal Intubation
Number analyzed (Participants) | 56 | 56
Participants | 22 | 35

2. Secondary Outcome: The Number of Participants With Severe Epistaxis
Description: The number of participants with severe epistaxis within 5 minutes following nasal tube placement.
Time Frame: Within 5 minutes following nasal intubation
Population: The number of patients with severe epistaxis in the use of the red rubber catheter vs. the standard insertion catheter
Measure: Count of Participants; unit: Participants
Arm/Group | Red Rubber Catheter Group | Standard Nasal Tracheal Intubation
Number analyzed (Participants) | 56 | 56
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Post-operative 24 hrs.
Arm/Group | Red Rubber Catheter Group | Standard Nasal Tracheal Intubation
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT03779984/Prot_SAP_ICF_000.pdf